CLINICAL TRIAL: NCT00546689
Title: Phase 1 Correlation Between Intestinal Parasites and Serum Level of Eosinophils and IgE in Individuals With HIV or AIDS
Brief Title: Correlation Between Intestinal Parasites and Serum Level of Eosinophils and IgE in Individuals With HIV or AIDS
Status: Completed | Type: Observational
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Other Study IDs: upeclin/HC/FMB-Unesp-02; Botucatu Medical School UNESP
Record Dates: First submitted 2007-10-18; First posted 2007-10-19 (Estimated); Last update posted 2008-04-18 (Estimated); Status verified 2007-10

CONDITIONS: HIV Infections
Keywords: HIV; aids; intestinal parasites; eosinophils; immunoglobulins; HIV/aids; Treatment Experienced
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; Intestinal Diseases, Parasitic

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Sample of Blood Sample of Feces
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1 , 2: those with HIV

SUMMARY:
Correlation between intestinal parasites and serum level of eosinophils and IgE in individuals with HIV or aids attended at clinical hospital of the Botucatu Medical School-UNESP

DETAILED DESCRIPTION:
The present study correlates intestinal parasitism and levels of eosonophils and of serum IgEs in patients attended at the C.H. of the School of Medicine - Botucatu/UNESP. Thirty adult patients with AIDS were analyzed in the use of HAART, aged 42 ±11 years, 14 (46.7%) male, excluding those that had used anthelminthics 30 days prior to collection. Socioeconomic questionaires were applied and 3 samples of feces were taken for parasitological exams (TF-test® method) and 5 ml of blood for counting eosinophils (automated hematological counter, Pentra 80, ABX) and IgE doses (equipment BN-100, Dade-Behring). The index of parasites was 10%, with E.nana (3.3%), E.coli (3.3%) and B.hominis (3.3%). Parasitized individuals were from an urban region with complete basic sanitation and good socioeconomic level. Normal eosinphil values were found in all samples and increased IgE values in 1 (33.3%) sample. The index of parasites was low due to good socioeconomic level and disease control. Augmented IgE levels corroborate the literature, which reports an increase characteristic of immune response in the face of parasitic infections in individuals with HIV or AIDS. In conclusion, new studies should be undertaken to evaluate the level of eosinophils associated with cytokines to obtain a better understanding of this correlation.

ELIGIBILITY:
Inclusion Criteria:

* HIV or AIDS
* age same or superior to 18 years,
* both sexes
* assisted by the Hospital of the Clinics of Botucatu Medical School-UNESP

Exclusion Criteria:

* use of anthelminthic in the period of 30 days antecedents the it dates from collection
* individuals that don't have all of the necessary evaluations to the objectives of the study
* individuals that abandon the attendance, or that you/they are to death during the study

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2007-03; Study Completion 2007-08 (Actual)

PRIMARY OUTCOMES:
all | one year

SECONDARY OUTCOMES:
all | one year

CONTACTS AND LOCATIONS:
Overall Officials: Paulo C Pereira, Phd, Study Chair — Botucatu Medical School - UNESP